CLINICAL TRIAL: NCT03753711
Title: Paraspinal Muscle Remodeling in Patients With Unilateral Lumbar Disc Herniation
Brief Title: Paraspinal Muscle Remodeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, Frank Vandenabeele, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LDH-UH
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Lumbar Disc Herniation
Keywords: lumbar disc herniation; hernia
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDH (lumbar disc hernia) (Experimental)
  Interventions: Procedure: Multifidus muscle biopsy during minimally invasive back surgery

INTERVENTIONS:
Procedure: Multifidus muscle biopsy during minimally invasive back surgery — Bilateral biopsy of the multifidus muscle in patient with a unilateral disc hernia.

SUMMARY:
Lumbar disc herniation is the most common diagnosed degenerative pathology in the lumbar spine with a prevalence of 2 to 3% in the adult population. Unilateral lumbar disc herniation is characterized by compression or irritation of the lumbar nerve roots or dural sac by either protrusion, extrusion or sequestration of the nucleus pulposus, mostly in the posterolateral region. Compression or irritation of the lumbar nerve roots and dural sac can induce unilateral sensory and motor symptoms. Therefore, it is the principal cause of lumbar spinal surgery.

Different imaging studies have investigated asymmetry of the paraspinal muscles in patient with unilateral low back pain due to lumbar discus herniation. Both animal and human studies indicate a reduction in total muscle cross-sectional area, increased fat infiltration and fibrosis within the lumbar multifidus at the affected side.

Increased fat infiltration is clinically important because there is a correlation between the amount of intramuscular fat and lumbar muscle dysfunction. Not only fat infiltration correlates with lumbar dysfunction, also a lower multifidus cross-sectional area is associated with and predictive for low back pain. This indicates that there is an association between paraspinal muscle changes/ remodeling and muscle dysfunction that could lead to low back pain.

The aim of this research is to quantify the decrease in muscle and muscle fibre size, the amount of fat infiltration, and the amount of fibrosis present within the multifidus muscle at the herniated side in relation to the unaffected side. The second aim is to investigate the possible role of different cell types in the process of muscle remodeling. The last aim of this study is to correlate these muscular changes with long-term functional outcomes such as pain, fear and disability. This information can possibly contribute to the etiology of paraspinal muscle changes, and provide a handgrip to future research.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lumbar disc hernia (diagnosed using MRI)
* Age between 18-55
* Understanding the Dutch language

Exclusion Criteria:

* Spinal surgery within the last year
* Degenerative or other spinal pathology (except disc hernia)
* Contraindications to undergo a MRI
* Other known pathologies that might affect muscle biology/ morphology

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
muscle biopsy sample (musculus multifidus) | day 1
  Histochemical analyses: Masson's trichrome and haematoxylin and eosin staining will be used to visualize connective and adipose tissues within a muscle cross-section.
muscle biopsy sample (musculus multifidus) | day 1
  Immunofluorescent analyses: Primary and secondary immunofluorescent antibody's against MHC I, IIA and IIX, laminin, satellite cells / muscle stem cells (PAX-7, MyoD, Myogenin), fibro-adipogenic cells/ mesenchymal progenitor cells (PDGFR-alfa) and myonuclei (DAPI) will be used.
muscle biopsy sample (musculus multifidus) | day 1
  Real-time PCR: Inflammatory markers and growth factors will be measured using real-time polymerase chain reaction.
MRI | day 1
  Medical imaging: Pre-operative MRI images will be requested from the department of radiology to measure total muscle cross-sectional area and intramuscular fat infiltration.

SECONDARY OUTCOMES:
Numeric Pain Rating Score (NPRS) | day 1
  this is a tool to provide an indication of the amount of pain a participant is feeling. It's a scale with 11 scores (0-10). It's a scale in which score 0 means 'no pain' and score 10 means 'the highest imaginable pain'. An improvement of 2 levels is considered clinically relevant.
Numeric Pain Rating Score (NPRS) | week 6
  this is a tool to provide an indication of the amount of pain a participant is feeling. It's a scale with 11 scores (0-10). It's a scale in which score 0 means 'no pain' and score 10 means 'the highest imaginable pain'. An improvement of 2 levels is considered clinically relevant.
Numeric Pain Rating Score (NPRS) | month 6
  this is a tool to provide an indication of the amount of pain a participant is feeling. It's a scale with 11 scores (0-10). It's a scale in which score 0 means 'no pain' and score 10 means 'the highest imaginable pain'. An improvement of 2 levels is considered clinically relevant.
Modified Oswestry Disability Index (ODI) | day1
  this is a questionnaire than has been proven valid and reliable to evaluate the restrictions that people with low back pain experience during their daily living. It consist of 10 items that will be scored on a 5 point scale. Using the total score you can calculate a percentage restriction degree. The score is calculated using the sum of the scores (0-5) from all 10 questions and multiply them times two. The final score is interpreted as following: 0-20%: minimal disability, 21-40%: moderate disability, 41-60%: severe disability, 61-80%: crippled, 81-100% bed bound.
Modified Oswestry Disability Index (ODI) | week 6
  this is a questionnaire than has been proven valid and reliable to evaluate the restrictions that people with low back pain experience during their daily living. It consist of 10 items that will be scored on a 5 point scale. Using the total score you can calculate a percentage restriction degree. The score is calculated using the sum of the scores (0-5) from all 10 questions and multiply them times two. The final score is interpreted as following: 0-20%: minimal disability, 21-40%: moderate disability, 41-60%: severe disability, 61-80%: crippled, 81-100% bed bound.
Modified Oswestry Disability Index (ODI) | month 6
  this is a questionnaire than has been proven valid and reliable to evaluate the restrictions that people with low back pain experience during their daily living. It consist of 10 items that will be scored on a 5 point scale. Using the total score you can calculate a percentage restriction degree. The score is calculated using the sum of the scores (0-5) from all 10 questions and multiply them times two. The final score is interpreted as following: 0-20%: minimal disability, 21-40%: moderate disability, 41-60%: severe disability, 61-80%: crippled, 81-100% bed bound.
Tampa Scale for Kinesiophobia (TSK) | day 1
  this is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. A higher score relates to more pain-related fear. A score >37/68 (with 68 being the highest possible score) means there is fear of movement present.
Tampa Scale for Kinesiophobia (TSK) | week 6
  this is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. A higher score relates to more pain-related fear. A score >37/68 (with 68 being the highest possible score) means there is fear of movement present.
Tampa Scale for Kinesiophobia (TSK) | month 6
  this is an ordinal 17 item questionnaire that inventories pain-related fear of movement for persons with subacute and chronic low back pain or fibromyalgia. A higher score relates to more pain-related fear. A score >37/68 (with 68 being the highest possible score) means there is fear of movement present.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandenabeele, prof. dr., Principal Investigator — Hasselt University; Sjoerd Stevens, drs., Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium